CLINICAL TRIAL: NCT02618616
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Group Study to Determine the Efficacy, Safety and Tolerability of Once Daily Oral ZPL-3893787- 18 (30 mg) Administered for 12 Weeks in Adult Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Determine the Efficacy of ZPL-3893787 in Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ziarco Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZPL389/102
Record Dates: First submitted 2015-11-27; First posted 2015-12-01 (Estimated); Results first posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ZPL-389 (Experimental): Each subject was given 30 mg ZPL-3893787 capsules, to be taken orally once daily (OD) for 12 weeks.
  Interventions: Drug: ZPL-3893787
- Placebo (Placebo Comparator): Each subject was given 30 mg capsules of matching placebo, to be taken orally OD for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZPL-3893787
  Other Names: ZPL389
  Arms: ZPL-389
Drug: Placebo
  Arms: Placebo

SUMMARY:
This was a randomized, double blind, placebo controlled, parallel group study in 129 subjects with moderate to severe psoriasis with a PASI score of at least 10. Following run-in, subjects were randomized and received either oral 30 mg ZPL-3893787 once daily or placebo once daily for 12 weeks.

DETAILED DESCRIPTION:
This was a randomized, double blind, placebo controlled, parallel group study in 129 subjects with moderate to severe psoriasis with a Psoriasis Area and Severity Index (PASI) score of at least 10 and an Investigator's Global Assessment (IGA) of 3 (0-4 scale). Following run-in subjects received either oral 30 mg ZPL-3893787 once daily or placebo once daily for 12 weeks. Subjects attended the clinic at Baseline (Day 0) when they were reviewed and confirmed they met inclusion/exclusion criteria. Subjects were then randomized and received either oral 30 mg ZPL-3893787 once daily or placebo once daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A documented history of moderate to severe plaque psoriasis for at least 6 months prior to screening.
* Male or female, aged ≥18 years.
* Psoriasis Area and Severity Index (PASI) ≥10 at both Screening and Day 0.
* An Investigator's Global Assessment (IGA) score ≥ 3 at both Screening and Day 0.
* Psoriasis affecting ≥10% body surface area (BSA) at Screening and Day 0.

Exclusion Criteria:

* Current diagnosis of Pustular, Guttate, Erythrodermic, exfoliative or only nail psoriasis or a diagnosis of inverse psoriasis without having plaque psoriasis.
* Concurrent skin disease (e.g. acne) of such severity in the study area that it could interfere with the study evaluation or presence of skin comorbidities that may interfere with study assessments.
* Active skin infections (e.g. impetigo, abscesses) or any other clinically apparent infections.
* Biologic treatments for psoriasis (e.g. Enbrel, Humira, Stelara, Cosentyx) within 3 months of the start of the Run-In.
* Phototherapy (e.g. UVA, UVB, PUVA) within 4 weeks of the start of the Run-In.
* Oral calcineurin inhibitors and immunosuppressants (e.g. cyclosporine, azathioprine, methotrexate) within 4 weeks of the start of the Run-In.
* Systemic corticosteroids within 4 weeks of the start of the Run-In.
* Oral antihistamines and leukotriene inhibitors and tricyclic antidepressants within 1 week of the start of the Run-In.
* Topical steroids (any potency), topical calcineurin inhibitors (tacrolimus, pimecrolimus), salicylic acid and urea containing treatments and coaltar preparations, topical and oral retinoids and vitamin D derivatives, within 1 week of the start of the Run-In.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Novartis
Locations (21):
- Belgium (4):
  - Belgium Study Centre, Brussels
  - Belgium Study Centre, Ghent
  - Belgium Study Centre, Leuven
  - Belgium Study Centre, Liège
- Germany (6):
  - German Study Centre, Berlin
  - German Study Centre, Goch
  - German Study Centre, Hamburg
  - German Study Centre, Hanover
  - German Study Centre, Mainz
  - German Study Centre, Münster
- Poland (7):
  - Polish Study Centre, Bialystok
  - Polish Study Centre, Gdansk
  - Polish Study Centre, Lodz
  - Polish Study Centre, Lublin
  - Polish Study Centre, Poznan
  - Polish Study Centre, Tarnów
  - Polish Study Centre, Wroclaw
- United Kingdom (4):
  - UK Study Centre, Blackpool
  - UK Study Centre, Bridgetown
  - UK Study Centre, Leeds
  - UK Study Centre, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each subject had a screening visit to confirm suitability to enter the study, followed by 7-day run-in period.
Period: Overall Study
Arm/Group | ZPL-389 | Placebo
Started | 87 | 42
Completed | 66 | 35
Not Completed | 21 | 7
Not completed — Lack of Efficacy | 4 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Adverse Event | 8 | 0
Not completed — Failure to comply with dosing/evaluation | 1 | 0
Not completed — Consent withdrawn by subject | 8 | 5
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): All randomized subjects who received at least one dose of study treatment.
Groups:
- ZPL-389: Each subject was given 30 mg ZPL-3893787 capsules, to be taken orally OD for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | ZPL-389 | Placebo | Total
Number analyzed (Participants) | 87 | 42 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (13.82) | 43.2 (12.64) | 44.1 (13.41)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 33 | 15 | 48
  Male | 54 | 27 | 81
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.24 (3.494) | 27.86 (3.575) | 28.12 (3.509)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Psoriasis Assessment of Severity Index (PASI) at Week 12
Description: The PASI is an assessment routinely used for evaluating and grading the severity of psoriatic lesions and their response to therapy. PASI divides the body into 4 regions: the head, trunk, upper extremities (arms) and lower extremities (legs). Each of these areas is assessed separately for erythema, in duration and scaling; these symptoms are scored on a 5-point scale from 0-4, where 0 = no symptoms and 4 =very marked. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 75 response represents a reduction of at least 75% from baseline in the PASI score.
Time Frame: From baseline to week 12
Population: Full analysis set (FAS): All randomized subjects who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | ZPL-389 | Placebo
Number analyzed (Participants) | 87 | 42
percentage change | -28.043 (38.4436) | -37.361 (32.3581)
Statistical Analysis 1: Comparison: ZPL-389 vs Placebo; ANCOVA of PASI at Week 12; Test type: Other; p = 0.8495, ANCOVA — The 1-sided p-value tests if the ZPL-389 Least square (LS) mean is < the placebo LS mean; least square difference = 8.7, 90% CI 1-sided [lower limit 8.4]

2. Secondary Outcome: PASI-50 and PASI-75 Responders at Week 12
Description: PASI-75 and PASI-50 are defined as a 75% and 50% reduction, respectively, from baseline in PASI score at Week 12.
Time Frame: From baseline to week 12
Population: FAS: All randomized subjects who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | ZPL-389 | Placebo
Number analyzed (Participants) | 87 | 42
Participants
  PASI-50 | 21 | 15
  PASI-75 | 12 | 6
Statistical Analysis 1: Comparison: ZPL-389 vs Placebo; Logistic Regression PASI-50; Test type: Other; p = 0.9058, Regression, Logistic; Odds Ratio (OR) = 0.562, 90% CI 2-sided [0.27 to 1.16]
Statistical Analysis 2: Comparison: ZPL-389 vs Placebo; Logistic Regression PASI-75; Test type: Other; p = 0.5422, Regression, Logistic; Odds Ratio (OR) = 0.946, 90% CI 2-sided [0.4 to 2.25]

3. Secondary Outcome: Improvement in Investigator Global Assessment (IGA) at Week 12
Description: An overall assessment of the severity of psoriasis was made, by the investigator, using the IGA at each visit. IGA scores take values on a 5-point scale from 0-4, where 0 = clear to 4 = severe disease. Responder is defined as a score of clear or almost clear, or a reduction of ≥2 levels. Success is defined as a score of clear or almost clear. Subjects with discontinued and missing data categories at Week 12 were considered non-responders.
Time Frame: From baseline to week 12
Population: FAS: All randomized subjects who received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | ZPL-389 | Placebo
Number analyzed (Participants) | 87 | 42
participants
  Responder | 10 | 6
  Success | 7 | 3

4. Secondary Outcome: Change From Baseline in the Numerical Rating Scale (NRS) for Pruritus (Worst Itch) at Week 12
Description: The pruritus NRS is an assessment tool used to assess the subject's worst itch as a result of psoriasis in the last 12 hours. The subjects completed the NRS each morning on (or soon after) rising and evening prior to retiring to bed. The subjects completed the NRS each morning on (or soon after) rising and evening prior to retiring to bed. They were asked the following question: On a scale of 0 (no itching) to 10 (itching as bad as you can imagine), please rate the worst itching that you felt over the last 12 hours.
Time Frame: From baseline to week 12
Population: FAS: All randomized subjects who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | ZPL-389 | Placebo
Number analyzed (Participants) | 87 | 42
percent change | -1.40 (2.659) | -1.78 (2.810)

5. Secondary Outcome: Patient Global Impression of Change (PGIC) a Week 12
Description: At the end of treatment (Week 12) or early termination visit, the subject was asked to rate their degree of improvement (or worsening) of their psoriasis compared to before the start of treatment with study drug, using a 7-point scale, standardized PGIC.
  Since the start of the study (dosing), my overall status is:
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Much worse
  7. Very much worse
Time Frame: From baseline to week 12
Population: FAS: All randomized subjects who received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | ZPL-389 | Placebo
Number analyzed (Participants) | 87 | 42
participants
  Very much improved | 12 | 3
  Much improved | 14 | 9
  Minimally improved | 22 | 11
  No change | 15 | 7
  Minimally worse | 5 | 3
  Much worse | 7 | 6
  Very much worse | 8 | 1
  Missing | 4 | 2

6. Secondary Outcome: Change From Baseline in Body Surface Area (BSA) and Percentage Change From Baseline at Week 12
Description: Assessment of the percentage of a subject's BSA affected by psoriasis was made by best estimates of the investigator at each visit. Hand-size measurement was considered to be the "best estimate" to measure the BSA by the investigators.
Time Frame: From baseline to week 12
Population: FAS: All randomized subjects who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | ZPL-389 | Placebo
Number analyzed (Participants) | 87 | 42
percentage of BSA | -2.8 (10.77) | -4.2 (9.62)

7. Secondary Outcome: Change From Baseline in the Daytime and Night Time NRS for Pruritus (Worst Itch) at Week 12
Description: The subjects completed the NRS each morning on (or soon after) rising and evening prior to retiring to bed. They were asked the following question: On a scale of 0 (no itching) to 10 (itching as bad as you can imagine), please rate the worst itching that you felt over the last 12 hours.
Time Frame: From baseline to week 12
Population: FAS: All randomized subjects who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ZPL-389 | Placebo
Number analyzed (Participants) | 87 | 42
score on a scale
  NRS for pruritus (daytime) at baseline | 4.32 (2.251) | 4.52 (2.748)
  Change in baseline at Week 12 (daytime): number analyzed (Participants) | 63 | 33
  Change in baseline at Week 12 (daytime) | -1.40 (2.765) | -1.42 (2.779)
  NRS for pruritus (night time) at baseline | 4.19 (2.299) | 4.34 (2.682)
  Change in baseline at Week 12 (night time): number analyzed (Participants) | 63 | 33
  Change in baseline at Week 12 (night time) | -1.35 (2.856) | -1.31 (2.860)

8. Secondary Outcome: Change From Baseline in the NRS for Sleep Disturbance at Week 12
Description: In the morning subjects were asked the following question to determine the level of sleep disturbance due to itching: On a scale of 0 (no sleep disturbance) to 10 (awake all night), please rate how much your sleep was disturbed by itch last night.
Time Frame: From baseline to week 12
Population: FAS: All randomized subjects who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ZPL-389 | Placebo
Number analyzed (Participants) | 87 | 42
score on a scale
  NRS for pruritus (sleep disturbance) at baseline | 2.48 (2.172) | 2.74 (2.559)
  Change in baseline at Week 12 (sleep disturbance): number analyzed (Participants) | 63 | 33
  Change in baseline at Week 12 (sleep disturbance) | -0.88 (2.417) | -0.93 (2.098)

9. Secondary Outcome: Change From Baseline in Total, Daytime and Night Time Duration of Itching at Week 12
Description: Subjects were asked the following question to determine their duration of itching: Over the last 12 hours approximately how many hours, if any, did you itch?
Time Frame: From baseline to week 12
Population: FAS: All randomized subjects who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ZPL-389 | Placebo
Number analyzed (Participants) | 87 | 42
hours
  Total duration of itching- Baseline | 5.74 (4.608) | 6.68 (5.637)
  Total duration of itching- Change at week 12: number analyzed (Participants) | 63 | 32
  Total duration of itching- Change at week 12 | -1.15 (4.525) | -1.16 (5.543)
  Daytime duration of itching-Baseline | 3.16 (2.682) | 3.57 (2.994)
  Daytime duration of itching-Change at week 12: number analyzed (Participants) | 63 | 32
  Daytime duration of itching-Change at week 12 | -0.60 (2.399) | 3.63 (3.034)
  Night time duration of itching-Baseline | 2.58 (2.072) | 3.11 (2.720)
  Night time duration of itching-Change at week 12: number analyzed (Participants) | 63 | 32
  Night time duration of itching-Change at week 12 | -0.55 (2.188) | -0.43 (2.581)

10. Secondary Outcome: Number of Participants for Each Verbal Rating Scale (VRS) Score for Pruritus at Week 12
Description: Subjects were asked to rate their itch over the last 12 hours using a list of adjectives describing different levels of symptom intensity: Over the last 12 hours how would you rate your itch? No itch; Mild; Moderate and Severe; Pruritus was evaluated by the subject, using the eDiary, twice daily for 1 week prior to the start of study treatment (run-in period) and during treatment (baseline to Day 84).
Time Frame: From baseline to week 12
Population: FAS: All randomized subjects who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | ZPL-389 | Placebo
Number analyzed (Participants) | 87 | 42
Participants
  Baseline - No itch | 2 | 2
  Baseline - Mild | 21 | 17
  Baseline - Moderate | 52 | 14
  Baseline - Severe | 12 | 9
  Week 12 - No itch | 17 | 11
  Week 12 - Mild | 19 | 10
  Week 12 - Moderate | 24 | 12
  Week 12 - Severe | 3 | 0
  Missing | 3 | 2
  Discontinued | 21 | 7

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 28 days post treatment up to maximum duration of 16 weeks
Description: Adverse events (AEs) are any untoward sign or symptom that occured during the study treatment
Arm/Group | ZPL-389 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/42
Serious Adverse Events (participants affected / at risk) | 5/87 | 0/42
Other Adverse Events (participants affected / at risk) | 26/87 | 6/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZPL-389 (N=87) | Placebo (N=42)
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZPL-389 (N=87) | Placebo (N=42)
Headache (Nervous system disorders) | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 11 | 1
Nasopharyngitis (Infections and infestations) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of the agreements with investigators may vary. However, the investigator is not prohibited from publishing. Any publications from a single site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.